CLINICAL TRIAL: NCT04605705
Title: NIRS: a Tool for the Diagnosis and Prevention of Acute Renal Failure in Pediatric Cardiac Surgery
Brief Title: NIRS for the Diagnosis and Prevention of Acute Renal Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Other Study IDs: FM389
Record Dates: First submitted 2020-03-16; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Renal Insufficiency, Acute
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood test for the dosage of creatinine and urea.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: NIRS values will be recorded during the surgery and until 24 hours postoperatively. No intervention will be done.
- Group 2: Several maneuvers will be performed in case the NIRS values are below 50%, such as an increase in cardiac output, temperature, hemoglobin to optimize the NIRS value by up to 80%.
  Interventions: Combination Product: Optimization of the cardiac output, the temperature, the hemoglobin in order to have the NIRS value by up to 80%.

INTERVENTIONS:
Combination Product: Optimization of the cardiac output, the temperature, the hemoglobin in order to have the NIRS value by up to 80%. — Several maneuvers will be performed in case the NIRS values are below 50%, such as an increase in cardiac output, temperature, hemoglobin to optimize the NIRS value by up to 80%.
  Groups: Group 2

SUMMARY:
This prospective study will take place at Hotel Dieu de France hospital in Lebanon. One hundred children undergoing cardiac surgery for congenital heart disease between May 2020 and May 2021 will be included. After obtaining the informed consent of the parents, demographic and surgical information will be collected. Serum creatinine, lactic acid, urinary neutrophil gelatinase-associated lipocalin marker (NGAL), and oxygen (O2) saturation will be measured before the operation.

A pediatric NIRS sensor will be placed on the right side below the costo-vertebral angle overlying the right kidney and continuous regional oxygen saturation (rSO2) will be recorded every 5 to 10 minutes throughout the operation until 24 hours after surgery. The children will be divided into 2 groups; 50 each. Grp 1: No clinical intervention was performed based on NIRS values. Grp 2: several maneuvers are performed such as an increase in cardiac output, temperature, hemoglobin to optimize the value of NIRS > 80%. All patients will receive standard standard care during the study period and continuous infusion of furosemide (0.5-1 mg / kg / 6 hours) within the first 24-48 hours postoperatively will be administered to all patients. Creatinine and lactic acid will be measured immediately postoperatively and then once a day until D2 and D7.

The urinary NGAL marker will be dosed immediately postoperatively and then at 2h, 6h, 12h and 24h with hourly monitoring of diuresis and NIRS until 24h postoperatively.

DETAILED DESCRIPTION:
This prospective study will take place at Hotel Dieu de France hospital in Lebanon. One hundred children aged 16 and under, undergoing cardiac surgery with cardiopulmonary bypass (CPB) for congenital heart diseases will be included between May 2020 and May 2021. The surgeries to be included will be the tetralogy of Fallot, transposition of the great arteries, ventricular septal defect, atrial septal defect and the atrioventricular canal defect. Any premature under 35 weeks of gestation, the presence of a genetic disease, an abnormal renal ultrasound, a preoperative renal failure with creatinine abnormal for age, or repeated urinary tract infections will be excluded from the study. After obtaining the informed consent of the parents, demographic information (age, weight, height, sex) will be collected..

Serum creatinine, lactic acid, urinary NGAL marker, and O2 saturation will be measured before the operation.

A pediatric NIRS sensor will be placed on the right side below the costo-vertebral angle covering the right kidney and continuous rSO2 will be recorded every 5 to 10 minutes throughout the operation as well as with each change of situation, then every hour in pediatric resuscitation until 24 hours postoperatively. The children will be divided into 2 groups of 50 patients each; Grp 1: No clinical intervention will be performed based on the NIRS and Grp 2: several maneuvers will be performed in case the NIRS values are below 50%, such as an increase in cardiac output, temperature, hemoglobin to optimize the NIRS value by up to 80%.

Surgical information (cardiac pathology, surgical procedure, operating time, duration of CPB, duration of aortic cross-clamping, duration of circulatory arrest, intraoperative complications) will be collected.

All patients will receive standard standard care during the study period. Patients will receive continuous infusion of furosemide (0.5-1 mg / kg / 6 hours) within the first 24-48 hours postoperatively.

Postoperatively, the need for catecholamines, the hemodynamic stability according to the Vasoactive-Inotropic Score (VIS), the delay to extubation, the stay in intensive care, the complications that occurred and the need for recourse to the dialysis will be noted.

Creatinine and lactic acid will be measured immediately postoperatively and then once a day until D2 and D7.

The urinary NGAL marker will be dosed immediately postoperatively and then at 2h, 6h, 12h and 24h with hourly monitoring of diuresis and NIRS until 24h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 16 years and under, undergoing cardiac surgery with cardiopulmonary bypass at the hotel Dieu de France Hospital, from September 2020 until September 2021.
* Surgeries to include: Tetralogy of Fallot, Transposition of great Vessels, ventricular septal defect, atrial septal defect and atrioventricular septal defect.
* Normal renal function
* Informed consent written and signed by the child's parents

Exclusion Criteria:

* The refusal of the patient's parents
* Patients with preoperative AKI
* Identification of renal or urinary anatomical abnormalities
* Premature infants <35 weeks of gestation
* Children with a known genetic or chromosomal abnormality
* Destination to a uni ventricular repair
* Repeated urinary tract infections before the surgery

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients aged 16 years and under, with normal renal function who are undergoing cardiac surgery with cardiopulmonary bypass from september 2020 until septembre 2021.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Impact of low renal NIRS values on renal function in children undergoing cardiac surgery. | 7 days
  Monitoring renal NIRS values during the surgery and until 24 hours in the ICU. All values are recorded. A dosage of creatinine is made upon arrival to the ICU , 24 hours later and one week later. A correlation between NIRS values and creatinine changes will be noticed.
Improving NIRS values prevent acute kidney injury in children undergoing cardiac surgery. | 7 days
  Optimizing renal NIRS values in children undergoing cardiac surgery. Each drop in NIRS values below 10% of its baseline is treated with transfusion and increasing the flow of CPB. Postoperatively, creatinine dosage is made upon arrival to the ICU, At day 1 and 7.

SECONDARY OUTCOMES:
Need for dialysis | 7 days
  Need for dialysis during the 1st week after the surgery
Duration of mechanical ventilation | 7 days
  Length of intubation and mechanical ventilation within the 1st postoperative week
Length of stay in intensive care units (ICU) | 1 month
  The length of stay in ICU within the 1st month after the surgery
Deaths within 30 days postoperative | 30 days
  Deaths within 30 days in children after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: AFRIDA GERGESS, M.D., Principal Investigator — Hotel Dieu de France Hospital
Locations (1):
- Hotel Dieu de France Hospital, Beirut, Lebanon